CLINICAL TRIAL: NCT01907386
Title: Abdominal Aortic Aneurysm Follow-up After Endovascular Repair by Non-invasive Vascular Elastography
Acronym: AAA-Elasto
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CE13.101
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2016-09

CONDITIONS: Aortic Aneurysm Abdominal; Endovascular Aneurysm Repair (EVAR)
Keywords: Endoleaks; Non-invasive vascular elastography
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- QSE-LSME and SSWI ultrasound (Other): QSE-LSME and SSWI ultrasound examinations combined with a clinically required CT-scan. We will screen 3 groups of 15 patients each, with at least one-year follow-up after EVAR, matched for sex, age and aneurysm diameter at baseline (before EVAR).
  Group 1. Patients without endoleak and a maximal diameter reduction at one year of at least 10% and a volume reduction of 20%.
  Group 2. Patients with a stable sac volume and diameter (less than 10% volume and 5% diameter variation within a year).
  Group 3. Patients with type I, type II or type V endoleak (endotension) with more than 10% diameter progression and 20% volume progression.
  Interventions: Other: QSE-LSME - SSWI Ultrasound

INTERVENTIONS:
Other: QSE-LSME - SSWI Ultrasound — Doppler ultrasound (DUS) and elastographic examinations will be performed using a single probe (6-1 MHz, Super Curved, Vermon, Tours, France) with the clinical Aixplorer system (Supersonic Imagine, Aix-en-Provence, France), a new generation ultrasound scanner providing an outstanding B-mode and color-Doppler image quality, allowing exportation of RF images for QSE-LSME acquisition and integrating the shear wave elastography (SSWI) mode.

SUMMARY:
Abdominal aortic aneurysm (AAA) is an abnormal dilatation of the aorta in the abdomen secondary to hypertension and atherosclerosis. Surgical treatment of AAA is increasingly being replaced by endovascular aneurysm repair (EVAR) using stent-grafts (SGs). However, the efficacy of this less invasive approach is often jeopardized by the incidence of persistent flow within the aneurysm, called endoleaks leading to aneurysm rupture if not properly detected and treated. Hence, a life long annual CT-scan surveillance is required increasing the cost of EVAR, exposing the patient to ionizing radiation and nephrotoxic contrast agent. The goal of this project is to adapt and test a new ultrasound technology called ultrasound elastography to improve patient follow-up after EVAR and ultimately avoid the use of CT-scans. This technique measures the deformation of the tissue secondary to blood pressure variation (quasi-static elastography) or to a shear wave generated by the ultrasound probe (dynamic elastography). The investigators will optimize 2 approaches to generate elastic maps of the AAA. One approach will be a quasi-static elastography (QSE-LSME) technique developed by our team giving an estimation of the deformation (strain) of the different components of the AAA by the blood pressure. The second is a dynamic elastography (SSWI) technique that will provide information on the elastic property of the AAA components.

DETAILED DESCRIPTION:
Experimental protocol: Optimization and validation of these 2 techniques will be completed in 3 experimental phases:

1. Preclinical validation: Abdominal aortic aneurysm and EVAR without endoleak (n=6), with a type I (n=6) and a type II (n=6) endoleak will be created in 18 mongrel dogs. QSE-LSME and SSWI acquisitions will be acquired before SG insertion and at 48H, 1, 3 months and at sacrifice at 6 months. The 2 techniques will be optimized to generate strain (QSE-LSME) and elasticity (SSWI) measurements of the simulated thrombus and vessel wall. CT-scan with prospective gating will be acquired on the AAA at least 6 different cardiac phases then segmented to allow 2D/3D registration of CT and elastographic acquisitions. Strain (QSE-LSME) and elasticity (SSWI) measurements of sac thrombus and vessel wall will be compared in the three experimental groups and correlated to sac pressure measurements, CT segmentation of sac components and pathologic evaluation.
2. Clinical feasibility, reproducibility and correlation with CT-angiography. From our EVAR database, 3 groups of 15 patients will be selected based on clinical and CT-angiography evolution. Group 1 will include patients without endoleak and AAA volume decrease of more than 20% following EVAR, group 2 patients without endoleak and no more than 10% sac volume variation and group 3 patients with endoleak or endotension and more than 20% sac volume increase. Ultrasound B-mode RF acquisitions with QSE-LSME and SSWI techniques will be acquired by two independent investigators. We will compare strain values of the different AAA components in the three groups. Thresholds will be tested to detect endoleak. Then strain values will be correlated with diameter, volume and stretch index variation between baseline and contemporary CT scans.
3. Prospective study validation of strain elasticity thresholds for endoleak detection and characterization of thrombus organization. The goal of this second clinical feasibility study is to collect longitudinal strain and elasticity measurements in the early post EVAR period (before one-year). We will include 15 patients with AAA scheduled for EVAR. These patients will have a baseline CT and baseline QSE-LSME and SSWI examination. Doppler ultrasound with QSE-LSME and SSWI examinations will then be performed at 3 and 12 months. The variation of strain and elastic values over time frames will be analyzed and correlated volume progression and endoleak occurrence on CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one-year follow-up after EVAR
* Willingness to comply with study follow-up requirements
* Written informed consent

Exclusion Criteria:

* Patients not clinically followed by CT-scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
QSE-LSME | Day 0: When the elastographic examinations (QSE-LSME, SSWI) and CT-scan will be completed
  We will compare strain values of the different AAA components in the three groups Then, we will test the best combination of strain criteria defined in the preclinical optimization and validation phase among three groups to evaluate if we can define a threshold to discriminate the 3 groups.
SSWI | Day 0: When the elastographic examinations (QSE-LSME, SSWI) and CT-scan will be completed
  Elasticity values of the aortic wall and thrombus in systolic and diastolic phase will be compared in the 3 groups

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Soulez, MD, M.Sc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada